CLINICAL TRIAL: NCT05832645
Title: A Randomized, Parallel Study Investigating the Effects of a Novel Approach to Mindfulness on Frequency and Duration of Meditation and Self-Reported Stress and Mood in Generally Healthy Adults
Brief Title: A Study Investigating the Effects of a Novel Mindfulness Approach on Frequency and Duration of Meditation and Self-Reported Stress and Mood in Generally Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otsuka Holdings Co., Ltd. (Industry)
Collaborators: Biofortis Innovation Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BIO-2304
Record Dates: First submitted 2023-04-13; First posted 2023-04-27 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior | interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A novel mindfulness approach (Experimental)
  Interventions: Other: Meditation with guided tea consumption
- Breathing meditation (Other)
  Interventions: Other: Breathing meditation

INTERVENTIONS:
Other: Meditation with guided tea consumption — Mindful consumption of tea along with an approximately 10-min guide
  Arms: A novel mindfulness approach
Other: Breathing meditation — 10-min breathing meditation
  Arms: Breathing meditation

SUMMARY:
The goal of this clinical trial is to compare the frequency and duration of meditation in generally healthy adults between:

1. A novel approach to mindfulness meditation encompassing guided tea consumption
2. Breathing meditation

Participants will be encouraged to meditate every day in either way listed above and asked to complete Daily Study Intervention Recall for 8 weeks.

Additionally, self-reported aspects of stress and mood will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 - 49 years (inclusive) at screening.
2. Born in the USA.
3. Self-report history of past participation in meditation but have not meditated in within 30 days (1 month) of screening.
4. Has an Apple ID, an email address linked to an Apple ID, and access to a dedicated smartphone capable of downloading and running the study specific app.
5. Able to download, install, and update apps using a smartphone.
6. Has access to hot water to prepare the tea beverage.
7. Regular (at least 3 days a week) consumer of caffeine.
8. Willing to maintain habitual diet (including supplements) and lifestyle (including avoidance of stressful events such as change in employment), physical activity patterns, and body weight during the study period.
9. Has no plan to change nicotine habits during the study period.
10. Has no health conditions that would prevent her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of the pre-screening questionnaire.
11. Understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Answered "Extremely" for all the positive feelings (energetic, lively, relaxed, and calm), or answered "Not at all" for all the negative feelings (lethargic, listless, irritated, and nervous), or gave same answer (e.g., Not at all) for all the feelings on the Mood State questionnaire completed during screening.
2. Visual or hearing impairments that cannot be corrected with glasses or contact lenses or hearing aids.
3. Self-reported taste or smell impairments within the past 30 days of screening.
4. Has a condition that prevents the subject from consuming caffeine (e.g., caffeine sensitivity, underlying heart condition).
5. Clinically diagnosed neurologic or psychiatric disorders (e.g., bipolar disorder, clinical depression, post-partum depression) currently requiring medication (such as antipsychotics, anticonvulsants, and antiparkinsonian agents as well as medications for bipolar disorder).
6. Clinically diagnosed sleep disorders (e.g., sleep apnea, insomnia, narcolepsy) requiring prescribed medical intervention (e.g., cognitive behavioral therapy, continuous positive airway pressure (CPAP), prescription medication such as zolpidem, zaleplon, eszopiclone, ramelteon, and suvorexant). Use of over-the-counter sleeping aid supplements such as melatonin, methylcobalamin (vitamin B12), 5-hydroxytryptophan (5-HTP), L-theanine, magnesium, and valerian is allowed.
7. Contraindication or allergy/sensitivity to any components in the study product or allergens present in the facility used to manufacture or pack the study product (see Appendix 10).
8. Elective hospitalizations planned (e.g., elective cosmetic procedures) during the study period.
9. Use of blood thinners (e.g., Warfarin).
10. Use of anti-hypertension medications.
11. Use of prescription stimulant medications [e.g., amphetamines/dextroamphetamine (Adderall), methylphenidate (Ritalin, Concerta), methamphetamine (Desoxyn), dextroamphetamine (Dexedrine), lisdexamfetamine (Vyvanse)]. Use of over-the-counter as-needed medications [e.g., for temporary pain relief (e.g., aspirin, ibuprofen, and acetaminophen), common cold/flu symptoms (pain relievers like aspirin, ibuprofen and acetaminophen; nasal decongestant sprays like oxymetazoline and phenylephrine; and oral decongestants, like pseudoephedrine), and seasonal allergies (e.g., Zyrtec, Claritin, Allegra)] is allowed.
12. Use of cannabis, marijuana or cannabinoid products, including those that are consumed, orally inhaled, smoked, applied topically, etc. within 6 months of screening.
13. Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. Subjects who are pregnant during the study will be discontinued.
14. Recent history of (within 12 months of screening) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
15. Has a condition the Clinical Investigator believes would interfere with her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
The frequency of meditation during the study | 8 weeks
  Frequency will be expressed as days whereby a meditation day is defined as a day where subjects completed at least one meditation session. Data will be obtained from the Daily Study Intervention Recall.
The total duration of time spent in meditation during the study | 8 weeks
  Data will be obtained from the Daily Study Intervention Recall.

SECONDARY OUTCOMES:
The average duration of time in meditation calculated weekly | weekly over 8 weeks
Changes from baseline (screening) in the total score of the Perceived Stress Scale | On Days 28 and 55
  Five-point scale from 0 (never) to 4 (very often). The total score ranges from 0 to 40 where higher values mean higher stress levels
Changes in the Mood Scale metrics | On Days 0 and 55
  * relaxed level
  * calm level
  * irritated level
  * focused level
  * anxious level
  * energetic level
  * lively level
  * lethargic level
  * listless level
  * nervous level
  * pleasure level (calculated)
  * arousal level (calculated)
  * vitality level (calculated)
  * stability level (calculated)
  The first ten items will be answered on a 6-point scale from 0 (not at all) to 5 (extremely). The last four metrics will be calculated according to the Two-Dimensional Mood Scale

OTHER OUTCOMES:
Survey related to meditation benefits | On Days 28 and 55
Product/Program Satisfaction Survey | On Days 0, 28 and 55

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis Innovation Services, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tanaka-Kanegae R, Yamada K, Cook CM, Blonquist TM, Taggart KD, Hamada K. Feasibility and Efficacy of a Novel Mindfulness App Used With Matcha Green Tea in Generally Healthy Adults: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2024 Dec 10;12:e63078. doi: 10.2196/63078. PMID 39657179